CLINICAL TRIAL: NCT04504929
Title: The Effectiveness of Dynamic Taping in Preventing Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: N201912094
Record Dates: First submitted 2020-06-22; First posted 2020-08-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2020-02

CONDITIONS: Fatigue; Muscle, Heart; Shoulder Pain; Sport Injury
MeSH Terms: conditions — Fatigue; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tape (Sham Comparator): participants received sham taping during pitching, and removed after pitching
  Interventions: Device: Sham tape
- Dynamic tape (Experimental): participants received dynamic taping during pitching, and removed after pitching
  Interventions: Device: Dynamic tape

INTERVENTIONS:
Device: Sham tape — Use sham type on the pitching shoulder
  Arms: Sham tape
Device: Dynamic tape — Use dynamic type on the pitching shoulder for supporting internal rotation
  Arms: Dynamic tape

SUMMARY:
The purpose of this study is to assess the efficacy of dynamic tape in prevent shoulder muscle fatigue.

DETAILED DESCRIPTION:
After being informed about the study and the potential of risk, all participants will undergo a screening to determine eligibility for study entry and giving written informed consent.

We will include 20 participants who have pitch 100 times with dynamic taping or shame taping in randomized sequence. There must be more than 2 weeks resting between 2 test. We will test maximal force in shoulder flexion, extension, abduction and adduction before and after test. We also record spins and speed of baseball for performance outcome.

To our hypothesis, we suggest dynamic taping could decrease the arm fatigue after long-term pitching.

ELIGIBILITY:
Inclusion Criteria:

* more than 20 years old
* amateur baseball player
* could tolerate pitching 100 times

Exclusion Criteria:

* shoulder pain who could not tolerate 100 pitching
* upper limb surgery history
* Allergy to topical agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in shoulder force after pitching | baseline and 2 weeks
  The dynamometer is a validated instrument assessing shoulder and arm force which is recorded in kilogram

SECONDARY OUTCOMES:
Change of pitching velocity during pitching | baseline and 2 weeks
  The speed dun is a validated instrument assessing pitching velocity which is recorded in kilometer per hour
Change of pitching spin rate during pitching | baseline and 2 weeks
  The STRIKE baseball is a new instrument assessing pitching spin rate and axis which is recorded in rate per minute
Change of delayed onset muscle soreness after pitching | baseline, 1 Day, 2 days, 3 days, 4 days, 5 days, 6 days, 7 days, 14 days
  Visual analog scale is a validated self-record measure to assess delayed onset muscle soreness, which score range is 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: YuHsaun Cheng, Master, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided